CLINICAL TRIAL: NCT05739409
Title: An Exploratory Clinical Study on the Safety and Efficacy of LILRB4 STAR-T Cells in the Treatment of Monocytic Leukemia
Brief Title: LILRB4 STAR-T Cell Therapy for Monocytic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022069
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Acute Myelogenous Leukemia; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LILRB4 STAR-T cells injection (Experimental): The study was divided into two phases: dose climbing and dose extension. Dose climbing stage: adopt the 3 + 3 dose climbing design principle, and the dose group is set as follows, in which, dose group-A is the backup dose reduction dose group, and dose group A is the starting dose:
  Dose Group-A: 3×105STAR+T cells / kg； Dose group A: 1×106STAR+T cells / kg； Dose group B: 3×106STAR+T cells / kg； Dose group C: 6×106STAR+T cells / kg； Dose group D: 1×107STAR+T cells / kg。
  Interventions: Biological: LILRB4 STAR-T cells injection

INTERVENTIONS:
Biological: LILRB4 STAR-T cells injection — The study population was relapsed/refractory acute myeloid leukemia and chronic myelomonocytic leukemia.Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of STAR-T cells. STAR-T cells will be intravenously infused with a escalated dose of 1E6#3E6#6E6#1E7 cells/kg

SUMMARY:
This is a single-center,single-arm,open-label phase I clinical study to determine the safety and efficacy of LILRB4 STAR-T cells in Monocytic Leukemia subjects.

DETAILED DESCRIPTION:
This study will recruit LILRB4-positive monocytic leukemia subjects who will receive cyclophosphamide and fludarabine on days -5 to -3 prior to cell infusion, followed by LILRB4 STAR-T cells. The primary objective of the study was to evaluate the safety and tolerability of LILRB4 STAR-T cells in subjects with monocytic leukemia. The secondary objective was to evaluate the therapeutic efficacy, pharmacodynamics and pharmacokinetics of LILRB4 STAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

-

1. Aged 18-70 years, gender is not limited 2. Acute myelogenous leukemia or chronic monocytic leukemia:

1. Subjects diagnosed with acute myelogenous leukemia according to WHO 2016 criteria and according to the "Chinese Guidelines for the Diagnosis and Treatment of Relapsed and Refractory Acute Myeloid Leukemia (2021 Edition)" should meet any of the following relapsed and refractory (R/R) acute myelogenous leukemia patients:

   1. Patients who have failed two cycles of standard chemotherapy;
   2. No remission was achieved after 1 cycle of the standard regimen and could not continue with the standard regimen due to age, comorbidities, physical status, and / or adverse risk factors;
   3. Relapse within 12 months after consolidation and intensification therapy after complete remission (CR);
   4. Relapse after 12 months but failed to respond to conventional treatment;
   5. two or more recurrences;
   6. persistent extramedullary leukemia;
   7. For age> 60 years: standard regimen chemotherapy due to age, comorbidities, physical status, and / or adverse risk factors, and treated with 4 cycles of demethylating drugs (such as decitabine and / or azacitidine) or 2 cycles of low-dose chemotherapy ± demethylating drugs。 Note: Definition of relapse: reoccurrence of leukemic cells in peripheral blood after CR or in bone marrow> 5% (except for other causes such as marrow regeneration after consolidation chemotherapy) or extramedullary infiltration of leukemic cells.
2. Chronic granule-monocytic leukemia (CMML) type 2 was diagnosed according to the World Health Organization (WHO) 2016 Hematopoietic and Lymphoid Tissue tumors and the Chinese Guidelines for the Diagnosis and Treatment of Chronic Grain-Monocytic Leukemia (2021 edition), and did not achieve remission after at least one treatment or relapsed after remission。 3. Eastern Cooperative Oncology Group physical status level is 0 to 2; 4. Bone marrow sample must be LILRB4 positive； 5. Major organs must meet the following criteria:

   1. Liver function: Total bilirubin≤1.5 times the upper limit of normal,glutamic-pyruvic transaminase and glutamic oxalacetic transaminase≤3 times the upper limit of normal,
   2. Renal function:Creatinine≤1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥60ml/min,
   3. Cardiac function:LVEF≥50%，
   4. Lung function:Defined as ≤grade 1 dyspnea and blood oxygen saturation >92%; 6. Female subjects of reproductive age or male subjects whose partners are women of reproductive age agree to use an effective method of contraception throughout the trial and for 12 months after cell infusion; 7. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Patients who have used chimeric antigen receptor T-cell immunotherapy therapy or any other gene transduction product within 3 months of signing the informed consent, except without detectable chimeric antigen receptor T-cell ratio or chimeric antigen receptor T-cell ratio below the lower test limit; or patients who have participated in other interventional clinical studies within 4 weeks prior to signing the informed consent；
2. Any of the following cardiovascular and cerebrovascular diseases occurred within 6 months before screening:

   1. congestive heart failure(NYHA stage III),myocardial infarction,unstable angina pectoris,congenital long QT syndrome,Anterior left block,coronary angioplasty,stent implantation,Coronary/peripheral artery bypass grafting,cerebrovascular accident,Transient ischemic attack or pulmonary embolism,Asymptomatic right bundle branch block was allowed;
   2. Serious arrhythmias requiring treatment (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes, etc.);
   3. uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg), a history of hypertensive crisis or hypertensive encephalopathy;
3. Subjects with positive hepatitis B surface antigen (HBsAg) or positive hepatitis B core antibody (HBcAb) and hepatitis B virus DNA copy number above the detection limit; subjects with positive hepatitis C virus (HCV) antibody and positive HCV RNA copy number above the detection limit; positive pallidum antibody test；
4. Patients with known systemic lupus erythematosus, combined active or uncontrolled autoimmune diseases (such as Crohns disease, rheumatoid arthritis, autoimmune hemolytic anemia, etc.), primary or secondary immune deficiency (such as HIV infection or severe infectious diseases, etc.)；
5. Previous or concurrent other incurable malignancies with unstable control,Affect the long-term survival of subjects, except for cured cervical carcinoma in situ, non-invasive basal cell or squamous cell skin cancer or other local prostate cancer after radical treatment, ductal carcinoma in situ after radical resection and at least 5 Years without recurrence of malignant tumor;
6. Patients with current disease or a previous history of central nervous system disease, such as seizures, stroke, severe brain injury, aphasia, paralysis, dementia, Parkinson's disease, mental illness, etc；
7. Patients living with an active central nervous system leukemia (CNSL)；
8. Patients who had prior solid organ transplantation or allogeneic hematopoietic stem cell transplantation (allo-HSCT) 6 months before screening；
9. Subjects with aGVHD and cGVHD at screening；
10. Subjects who have had any of the following drugs or treatments within the specified time period prior to apheresis:

    1. Administered any immunosuppressant within 2 weeks prior to apheresis;
    2. Received any chemotherapy within 2 weeks or 3 half-lives, whichever is shorter, prior to apheresis;
    3. Received any macromolecule or small molecule targeted therapy such as monoclonal antibody, antibody-drug conjugate (ADC), double antibody, etc. within 4 weeks before apheresis or within 3 half-lives (whichever is shorter);
11. Those with mental illness or history of drug abuse;
12. Pregnant or breastfeeding subjects;
13. The investigator believes that there are other factors that are not suitable for inclusion or that affect subjects participating in or completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability | 12 months
  Subjects are observed for dose-limiting toxicity(DLT) after LILRB4 STAR-T cells infusion, with the recording of adverse events(AE) and serious adverse events(SAE), with a focus on cytokine release syndrome(CRS) and immune cell-associated neurotoxicity(ICANS).All of the AE ratings were assessed according to the CTCAE.

SECONDARY OUTCOMES:
Antitumor efficacy | 12 months
  After infusion of LILRB4 STAR-T cells, the subjects underwent bone marrow puncture every month to evaluate the tumor load in the bone marrow. The efficacy evaluation included complete morphological remission, complete remission with incomplete recovery of blood cytology, and partial remission.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (2):
- China (2):
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No